CLINICAL TRIAL: NCT01722409
Title: Sevoflurane, Laryngeal Mask Airway and Single-dose Dexmedetomidine: A Better Choice for Patients Undergoing Endovascular Coil Embolization
Brief Title: A Better Choice for Patients Undergoing Endovascular Coil Embolization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Associate professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20121009
Record Dates: First submitted 2012-11-03; First posted 2012-11-06 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2013-10

CONDITIONS: Intracranial Aneurysms
Keywords: dexmedetomidine, endovascular coil embolization
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Sevoflurane; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sevoflurane and saline infusion (No Intervention): After induction of general anesthesia, Group S received a placebo infusion of normal saline.
- sevoflurane and 0.5 μg/kg dexmedetomidine (Experimental): After induction of general anesthesia, Group DEX1 received a single dexmedetomidine dose of 0.5 μg/kg over 10 minutes.
  Interventions: Drug: sevoflurane and 0.5 μg/kg dexmedetomidine
- sevoflurane and 1 μg/kg dexmedetomidine (Experimental): After induction of general anesthesia, Group DEX2 received a single dexmedetomidine dose of 1 μg/kg over 10 minutes.
  Interventions: Drug: sevoflurane and 1 μg/kg dexmedetomidine

INTERVENTIONS:
Drug: sevoflurane and 0.5 μg/kg dexmedetomidine — After induction of general anesthesia, Group DEX1 received a single dexmedetomidine dose of 0.5 μg/kg over 10 minutes.
  Other Names: DEX1
  Arms: sevoflurane and 0.5 μg/kg dexmedetomidine
Drug: sevoflurane and 1 μg/kg dexmedetomidine — After induction of general anesthesia, Group DEX2 received a single dexmedetomidine dose of 1 μg/kg over 10 minutes.
  Other Names: DEX2
  Arms: sevoflurane and 1 μg/kg dexmedetomidine

SUMMARY:
The investigators designed a double-blind, randomized placebo-controlled study to determine the effects of dexmedetomidine on the recovery characteristics of patients who were scheduled to undergo endovascular coil embolization.

ELIGIBILITY:
Inclusion Criteria:18-65 years old ASA I or ASA II patients undergoing ECE treatment for intracranial aneurysms were included.

Exclusion Criteria:Patients were excluded based on the following parameters: older than 65 yrs, a history of mental illness, recent use of sedatives or analgesics and with sensation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Observing the recovery characteristics of patients who were scheduled to undergo endovascular coil embolization. | At the end of the operation and 24 hours later
  The time from termination of the general anesthetic to the time that the patient's eyes opened. Anesthesiologists collected information on emergence agitation, postoperative nausea and vomiting for 24 hours after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, M.D.,PhD., Study Chair — Dept. of Anesthesiology, the First Hospital of CMU
Locations (1):
- Wen-fei Tan, Shenyang, Liaoning, China